CLINICAL TRIAL: NCT02634372
Title: Single-blind, Randomized Controlled Comparison of EMDR Versus Supportive Therapy in Affective Relapse Prevention in Bipolar Patients With a History of Trauma
Brief Title: EMDR vs Supportive Therapy in Relapse Prevention in Traumatized Bipolar Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FIDMAG Germanes Hospitalàries (Other)
Collaborators: Hospital Clinic of Barcelona (Other); Hospital del Mar (Other); Hospital Universitari de Bellvitge (Other); Instituto de Salud Carlos III (Other Government); Centro de Investigación Biomédica en Red de Salud Mental (Network)
Responsible Party: Principal Investigator, Benedikt Lorenz Amann, Senior Research fellow, FIDMAG Germanes Hospitalàries
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI15/02242
Record Dates: First submitted 2015-12-03; First posted 2015-12-18 (Estimated); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Traumatic event; Eye Movement Desensitization Reprocessing; Supportive therapy; Relapse prevention
MeSH Terms: conditions — Bipolar Disorder | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EMDR Therapy (Experimental): EMDR: 20 individual sessions 60 minutes each for 6 months
  Interventions: Behavioral: EMDR therapy
- Supportive therapy (Active Comparator): Supportive therapy: 20 individual sessions 60 minutes each for 6 months.
  Interventions: Behavioral: Supportive Therapy

INTERVENTIONS:
Behavioral: EMDR therapy — EMDR: We designed a specific EMDR Bipolar Protocol which consists of a detailed interview with respect to traumatic events, the treatment of those with the EMDR standard protocol, and five new specific bipolar adapted EMDR protocols focusing on adherence, insight, de-idealisation of manic symptoms, prodromal symptoms and moodstabilization.
  Arms: EMDR Therapy
Behavioral: Supportive Therapy — Supportive therapy: Therapists adopt a client-centred focus, meaning that whatever problems the patient presents will be dealt with by providing emotional support and general advise. If no specific topic is mentioned by the patient, information about bipolar disorder and medication will be delivered by the therapist without referring to written or any other material.
  Arms: Supportive therapy

SUMMARY:
The purpose of this study is to determine whether EMDR (vs supportive therapy) is effective in relapse prevention over an observational period of 2 years in bipolar patients with a history of traumatic events.

DETAILED DESCRIPTION:
Background:

The intervention strategies available for bipolar disorder are essentially pharmacotherapy and psychosocial interventions such as cognitive behavioral therapy, psychoeducation, and interpersonal and family therapy. However, despite the everyday use in clinical practice of both types of intervention, almost 70% of patients with bipolar disorder suffer an affective relapse within two years. Although the origin of this is multi-causal, an emerging research topic is the association of bipolar disorder with posttraumatic stress disorder (PTSD). Data from the STEP-BD study showed a prevalence of 20% of PTSD in a sample of 3158 bipolar patients, a rate almost three times higher than the prevalence of PTSD in the general population. This comorbidity has important clinical implications as the traumatized bipolar patients suffer from more rapid cycling, more suicide attempts, more substance abuse, have lower quality of life and more (hypo) manic and depressive symptoms than bipolar patients without PTSD. The results are similar in populations with severe mental illness and a history of trauma (not necessarily diagnosis of PTSD). These populations have more affective episodes, more psychiatric symptoms, increased risk of suicide, more frequency of risk sexual behaviors, more admissions to psychiatric hospitals and in overall, a greater risk of being re-traumatized.

The strength of the evidence supporting the clinically relevant effects of PTSD and/or history of trauma in bipolar disorder contrasts with a surprising lack of trials aimed at treating patients who have experienced traumatic events. One form of treatment that is being increasingly used in PTSD therapy is Eye Movement Desensitization and Reprocessing (EMDR). This integrative psychotherapeutical approach uses standardized protocols and elements of cognitive-behavioral, interpersonal, and body-centered therapies in conjunction with dual stimulation (e.g. horizontal eye movements from side to side). The results of two independent meta-analyzes have shown that the EMDR therapy is as effective in the treatment of PTSD symptoms as cognitive behavioral therapy. The treatment with EMDR has also been tested successfully versus exposition therapy and waiting list in a large randomized controlled trial in patients with psychosis and PTSD. Their results showed a significant reduction of trauma scores in both intervention in comparison to the waiting list and both intervention were regarded as safe with respect to exacerbation of psychotic symptoms. Our group carried out the first randomized controlled pilot study of EMDR in bipolar traumatized patients with subsyndromal symptomatology. Our results showed that the EMDR intervention not only reduced the symptoms associated with trauma in the patients, but also had beneficial effects on the symptoms of subsyndromal mood. Following the results this study, our research group has developed a specific and comprehensive EMDR protocol for bipolar patients with a history of trauma. This protocol consists of a comprehensive survey of traumatic events, the intervention and processing of these events according to the Shapiro standard protocol and 5 sub-protocols directed to (a) enhance treatment adherence, (b) increase insight, (c) treat prodromal symptoms, (d) work on the de-idealization of manic symptoms and (e) provide mental stabilization.

Aims and hypotheses:

The main objective of this study is to examine if EMDR therapy with protocols specific to bipolar patients with a history of traumatic events can act as a mood stabilizer. This would result in less affective relapses and better overall and cognitive functioning after 6 months of therapy in the group that received EMDR submit compared with the ST group. Other related aims of this project are to expand the available options for psychosocial intervention in bipolar disorder, to demonstrate that the EMDR therapy is a safe and effective tool in traumatized bipolar patients and that treatment with EMDR lead to an improvement in the course and prognosis of the disease.

Hypotheses:

1. The EMDR group will show less affective relapses at 12 and 24 months follow-up compared to the ST group.
2. Patients in the EMDR group will show less affective symptoms compared to the ST group at evaluations at 6, 12 and 24 months.
3. Patients in the EMDR group will show better cognition and functioning compared to the ST group at evaluations at 6, 12 and 24 months.

Design:

Single-blind randomized clinical trial (1:1) with two parallel branches, stratified by center for age, sex, number of previous affective episodes and cognitive state. The preventive effect of two psychological interventions, individual EMDR therapy or ST plus pharmacological treatment in patients diagnosed with bipolar I and II disorder with history of traumatic events, in a current affective phase of euthymia or subsyndromal symptoms will be evaluated. The comparative clinical effect in both branches of intervention will be assessed at five time points. There will be a pre-intervention baseline assessment, a post-intervention assessment at 6 months and follow-up evaluations at 12, 18 and 24 months.

Clinical and diagnostic variables:

1. Clinical diagnosis of the participants will employ DSM-IV-TR criteria.
2. Clinical Severity of the participants will be assessed by different instruments:

   1. Bipolar Depression Rating Scale (BDRS): The BDRS is the most up-to-date and appropriate tool to assess depressive and mixed symptoms in bipolar patients. Our group has been involved in the translation and validation of the scale into Spanish.
   2. Young Mania Rating Scale (YMRS) which is validated in Spanish: YMRS is a hetero-administered scale of composed of 11 items aimed at quantifying the severity of manic and hypo manic episodes.
   3. Clinical Global Impression Scale modified for bipolar disorder (CGI-BP-M), Spanish validation: The CGI-BP-M scale consists of 3 subscales; the first two assess the severity of acute symptoms of mania and depression, and the third evaluates the longitudinal severity of the disease. Each subscale has seven sub-categories with scores from 1 to 7 rating the severity of the disorder as normal, low, mild, moderate, marked, severe or very severe.

   Other clinical variables will be collected via the medical history of the patients and using a specific CRF for the study such as age of onset of the disorder, number of relapses, number of previous episodes, history and number of suicide attempts and pharmacological variables such as the number, type and dose of drugs.
3. Trauma symptoms, cognitive profiles and overall functioning will be evaluated by the following instruments:

   1. Clinician-Administered PTSD Scale (CAPS) which is validated in Spanish.
   2. Impact of Event Scale Revised (IES-R).
   3. Distressing Event Questionnaire.
   4. Traumatic Life Events Questionnaire.

   c. Functioning Assessment Short Test (FAST). d. Screen for Cognitive Impairment in Psychiatry (SCIP) which is validated in Spanish.

   e. Screen for social cognition, emotional intelligence: Mayer-Salovery-Caruso Emotional Intelligence Test.

   Statistical analysis:
   1. Computation of sample size The study will assess the relative efficacy of a specific EMDR intervention protocol versus Supportive Therapy (ST) in the clinical stabilization (decrease in the number of relapses) of traumatized bipolar patients. For this reason the number of affective episodes after treatment with a follow up of 24 months will be used as the dependent variable of the study. The sample size computation is based on a recent study comparing CBT versus ST with 24 months follow up on the relapse in bipolar patients. The calculation of the sample size was based on a survival analysis using the statistical package "powerSurvEpi" for R (http://www.r-project.org/) using an alpha = 0.005 instead of 0.05 for allow correction for multiple comparisons. The number of patients required to detect a hazard ratio = 2 in a cox regression with a statistical power of 80% and alpha = 0.005 is n = 36 per intervention group (two groups, EMDR and ST, equals to a total n = 72). A sample of this size should show clinically relevant differences. Assuming a percentage of drop-outs of about 10-15% of the participants it would be necessary to recruit approximately 82 patients, 41 allocated in each intervention arm.
   2. Analysis of the main variables The baseline distribution of socio-demographic and clinical characteristics between the groups will be analyzed using descriptive statistics. Continuous variables with a normal distribution will be analyzed with Multivariate Analysis of Variance (MANOVA). The main hypothesis of survival time (in weeks) will be analyzed using Kaplan-Meier curves with tests of significance tests based on log-rank test. The change in baseline clinical variables compared to baseline at strategic time points of the trial will be analyzed by repeated measures ANOVA factor in for time, treatment conditions and their interaction. The Wilcoxon test will be used in cases that do not meet the assumptions of normality. Between groups differences in main categorical and clinical variables will be analyzed using the Chi-squared test. Those variables that are statistically significant will be used as covariates in a linear logistic regression of factors associated with the magnitude of the effect in order to determine which factors are better predictors of performance. For each of the analyses the effect size index (Hedges g index or Pearson r index) will be estimated. The latest version of the SPSS software (v. 18, 20) will be used to carry out all the statistical analysis.
   3. Analysis of clinical efficacy The mains statistical analysis will employ an intention to treat (ITT) approach to provide unbiased comparisons among the treatment groups. The "Last Observation Carried Forward" approach (LOCF) will be employed as a measure of minimizing losses.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfill diagnosis of bipolar I or II disorder, following DSM-IV-RT criteria
* Outpatients
* History of 2 to 6 affective episodes in previous year
* Patients are included in the study 1) in euthymia, defined as Bipolar Depression Rating Scale (BDRS) <8 and Young Mania Rating Scale (YMRS) <8 or 2) with subsyndromal symptoms, defined as BDRS ≥8 and <14 and/or YMRS ≥8 and <12
* Patients suffered at least from one traumatic event, evaluated by the Distressing Event Scale, Traumatic Life Events Questionnaire, Impact of Event Scale and Subjects Units of Distress.

Exclusion Criteria:

* Neurological disease
* Currently in a manic phase (YMRS>18), mixed phase (BDRS≥10 in mixed subscale of BDRS, max.: 15) or depressive phase (BDRS >18)
* Acute suicidal plans
* Substance Use Disorder within last 3 months (except of nicotine abuse/dependency)
* Trauma focused therapy within last 12 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-03; Primary Completion 2022-03 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Number of depressive, hypomanic, manic or mixed episodes | Change of relapses from baseline to visits at 6, 12 and 24 months
  Affective relapses are defined as: Depressive relapse: score>18 in the BDRS, and a score>3 in the CGI-BP-M, depressive subscale. Hypomanic relapse: a YMRS score between 7 and 20, and a score of 3 or 4 in the CGI-BP-M, the manic subscale. Manic relapse: a YMRS score of >20, and the CGI-BP-M, the manic subscale, score>4. Mixed relapse: a BDRS score>10 in the mixed subscale (max. 15), and a score >4 in the CGI-BP-M, depressive and manic subscales.

SECONDARY OUTCOMES:
Depressive symptoms | Change from baseline in depressive symptoms at 3, 6, 12 and 24 months
  To measure changes in depressive symptoms we will use the BDRS, and the CGI-BP-M, the depressive subscale.
(Hypo)manic symptoms | Change from baseline in (hypo)manic symptoms at 3, 6, 12 and 24 months
  To measure changes in (hypo)manic symptoms we will use the YMRS and the CGI-BP-M, the manic subscale.
Mixed symptoms | Change from baseline in mixed symptoms at 3, 6, 12 and 24 months
  To measure changes in mixed symptoms we will use the YMRS, the BDRS (mixed subscale) and the CGI-BP-M, the depressive and manic subscale.
Trauma associated symptoms | Change from baseline in trauma symptoms at 3, 6, 12 and 24 months
  To measure changes in trauma associated symptoms, the CAPS, IES, TLEQ and DEQ will be used.
Functioning | Change from baseline in functioning at 3, 6, 12 and 24 months
  To measure changes in functioning the FAST will be used.
Cognitive impairment | Change from baseline in cognition at 3, 6, 12 and 24 months
  To measure changes in cognition the SCIP will be used.
Social cognition and emotional intelligence | Change from baseline in cognition at 3, 6, 12 and 24 months
  To measure changes in social cognition and emotional intelligence the MSCEIT will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Benedikt L Amann, MD, Principal Investigator — Institut Hospital del Mar d'Investigacions Mèdiques
Locations (1):
- Institut Hospital del Mar d'Investigacions Mèdiques, Barcelona, Spain

REFERENCES:
- [Background] Brackett MA, Salovey P. Measuring emotional intelligence with the Mayer-Salovery-Caruso Emotional Intelligence Test (MSCEIT). Psicothema. 2006;18 Suppl:34-41. PMID 17295955
- [Background] Pino O, Guilera G, Rojo JE, Gomez-Benito J, Bernardo M, Crespo-Facorro B, Cuesta MJ, Franco M, Martinez-Aran A, Segarra N, Tabares-Seisdedos R, Vieta E, Purdon SE, Diez T, Rejas J; Spanish Working Group in Cognitive Function. Spanish version of the Screen for Cognitive Impairment in Psychiatry (SCIP-S): psychometric properties of a brief scale for cognitive evaluation in schizophrenia. Schizophr Res. 2008 Feb;99(1-3):139-48. doi: 10.1016/j.schres.2007.09.012. Epub 2007 Oct 23. PMID 17959358
- [Background] Purdo SE: The Screen for Cognitive Impairment in Psychiatry (SCIP): Instructions and three alternate forms. PNLInc, Edmonton, Alberta, 2005.
- [Background] Reinares M, Sanchez-Moreno J, Fountoulakis KN. Psychosocial interventions in bipolar disorder: what, for whom, and when. J Affect Disord. 2014 Mar;156:46-55. doi: 10.1016/j.jad.2013.12.017. Epub 2013 Dec 25. PMID 24439829
- [Background] Simhandl C, Konig B, Amann BL. A prospective 4-year naturalistic follow-up of treatment and outcome of 300 bipolar I and II patients. J Clin Psychiatry. 2014 Mar;75(3):254-62; quiz 263. doi: 10.4088/JCP.13m08601. PMID 24717379
- [Background] Hernandez JM, Cordova MJ, Ruzek J, Reiser R, Gwizdowski IS, Suppes T, Ostacher MJ. Presentation and prevalence of PTSD in a bipolar disorder population: a STEP-BD examination. J Affect Disord. 2013 Sep 5;150(2):450-5. doi: 10.1016/j.jad.2013.04.038. Epub 2013 May 23. PMID 23706842
- [Background] Quarantini LC, Miranda-Scippa A, Nery-Fernandes F, Andrade-Nascimento M, Galvao-de-Almeida A, Guimaraes JL, Teles CA, Netto LR, Lira SB, de Oliveira IR, Post RM, Kapczinski F, Koenen KC. The impact of comorbid posttraumatic stress disorder on bipolar disorder patients. J Affect Disord. 2010 Jun;123(1-3):71-6. doi: 10.1016/j.jad.2009.08.005. Epub 2009 Sep 3. PMID 19732957
- [Background] Simhandl C, Radua J, Konig B, Amann BL. The prevalence and effect of life events in 222 bipolar I and II patients: a prospective, naturalistic 4 year follow-up study. J Affect Disord. 2015 Jan 1;170:166-71. doi: 10.1016/j.jad.2014.08.043. Epub 2014 Sep 6. PMID 25240845
- [Background] Mueser KT, Goodman LB, Trumbetta SL, Rosenberg SD, Osher fC, Vidaver R, Auciello P, Foy DW. Trauma and posttraumatic stress disorder in severe mental illness. J Consult Clin Psychol. 1998 Jun;66(3):493-9. doi: 10.1037//0022-006x.66.3.493. PMID 9642887
- [Background] McElroy SL. Diagnosing and treating comorbid (complicated) bipolar disorder. J Clin Psychiatry. 2004;65 Suppl 15:35-44. PMID 15554795
- [Background] Shapiro F. Eye movement desensitization: a new treatment for post-traumatic stress disorder. J Behav Ther Exp Psychiatry. 1989 Sep;20(3):211-7. doi: 10.1016/0005-7916(89)90025-6. PMID 2576656
- [Background] Bisson JI, Ehlers A, Matthews R, Pilling S, Richards D, Turner S. Psychological treatments for chronic post-traumatic stress disorder. Systematic review and meta-analysis. Br J Psychiatry. 2007 Feb;190:97-104. doi: 10.1192/bjp.bp.106.021402. PMID 17267924
- [Background] Seidler GH, Wagner FE. Comparing the efficacy of EMDR and trauma-focused cognitive-behavioral therapy in the treatment of PTSD: a meta-analytic study. Psychol Med. 2006 Nov;36(11):1515-22. doi: 10.1017/S0033291706007963. Epub 2006 Jun 2. PMID 16740177
- [Background] van den Berg DP, de Bont PA, van der Vleugel BM, de Roos C, de Jongh A, Van Minnen A, van der Gaag M. Prolonged exposure vs eye movement desensitization and reprocessing vs waiting list for posttraumatic stress disorder in patients with a psychotic disorder: a randomized clinical trial. JAMA Psychiatry. 2015 Mar;72(3):259-67. doi: 10.1001/jamapsychiatry.2014.2637. PMID 25607833
- [Background] Novo P, Landin-Romero R, Radua J, Vicens V, Fernandez I, Garcia F, Pomarol-Clotet E, McKenna PJ, Shapiro F, Amann BL. Eye movement desensitization and reprocessing therapy in subsyndromal bipolar patients with a history of traumatic events: a randomized, controlled pilot-study. Psychiatry Res. 2014 Sep 30;219(1):122-8. doi: 10.1016/j.psychres.2014.05.012. Epub 2014 May 15. PMID 24880581
- [Background] Amann BL, Batalla R, Blanch V, Capellades D, Carvajal MJ, Fernández I, García F, Lupo W, Ponte M, Sánchez J, Sanfiz J, Santed A and Luber M: The EMDR Therapy Protocol for Bipolar Disorder. In M. Luber (Ed.), Eye Movement Desensitization and Reprocessing (EMDR) Scripted Protocols and Summary Sheets: Treating trauma, anxiety and mood-related conditions. New York: Springer, 2015 (p 223-287).
- [Background] Berk M, Malhi GS, Cahill C, Carman AC, Hadzi-Pavlovic D, Hawkins MT, Tohen M, Mitchell PB. The Bipolar Depression Rating Scale (BDRS): its development, validation and utility. Bipolar Disord. 2007 Sep;9(6):571-9. doi: 10.1111/j.1399-5618.2007.00536.x. PMID 17845271
- [Background] Sarro S, Madre M, Fernandez-Corcuera P, Valenti M, Goikolea JM, Pomarol-Clotet E, Berk M, Amann BL. Transcultural adaption and validation of the Spanish version of the Bipolar Depression Rating Scale (BDRS-S). J Affect Disord. 2015 Feb 1;172:110-5. doi: 10.1016/j.jad.2014.10.009. Epub 2014 Oct 12. PMID 25451403
- [Background] Young RC, Biggs JT, Ziegler VE, Meyer DA. A rating scale for mania: reliability, validity and sensitivity. Br J Psychiatry. 1978 Nov;133:429-35. doi: 10.1192/bjp.133.5.429. PMID 728692
- [Background] Colom F, Vieta E, Martinez-Aran A, Garcia-Garcia M, Reinares M, Torrent C, Goikolea JM, Banus S, Salamero M. [Spanish version of a scale for the assessment of mania: validity and reliability of the Young Mania Rating Scale]. Med Clin (Barc). 2002 Sep 28;119(10):366-71. doi: 10.1016/s0025-7753(02)73419-2. Spanish. PMID 12372167
- [Background] Vieta Pascual E, Torrent Font C, Martinez-Aran A, Colom Victoriano F, Reinares Gabnepen M, Benabarre Hernandez A, Comes Forastero M, Goikolea Alberdi JM. [A user-friendly scale for the short and long term outcome of bipolar disorder: the CGI-BP-M]. Actas Esp Psiquiatr. 2002 Sep-Oct;30(5):301-4. Spanish. PMID 12372226
- [Background] Blake DD, Weathers FW, Nagy LM, Kaloupek DG, Gusman FD, Charney DS, Keane TM. The development of a Clinician-Administered PTSD Scale. J Trauma Stress. 1995 Jan;8(1):75-90. doi: 10.1007/BF02105408. PMID 7712061
- [Background] Bobes J, Calcedo-Barba A, Garcia M, Francois M, Rico-Villademoros F, Gonzalez MP, Bascaran MT, Bousono M; Grupo Espanol de Trabajo para el Estudio del Trastornostres Postraumatico. [Evaluation of the psychometric properties of the Spanish version of 5 questionnaires for the evaluation of post-traumatic stress syndrome]. Actas Esp Psiquiatr. 2000 Jul-Aug;28(4):207-18. Spanish. PMID 11116791
- [Background] Weiss DS, Marmar CR. The Impact of Event Scale - Revised, Assessing Psychological Trauma and PTSD. Guilford Press, New York, 1997 pp.399-411
- [Background] Kubany ES, Leisen MB, Kaplan AS, Kelly MP. Validation of a brief measure of posttraumatic stress disorder: the Distressing Event Questionnaire (DEQ). Psychol Assess. 2000 Jun;12(2):197-209. doi: 10.1037//1040-3590.12.2.197. PMID 10887766
- [Background] Kubany ES, Haynes SN, Leisen MB, Owens JA, Kaplan AS, Watson SB, Burns K. Development and preliminary validation of a brief broad-spectrum measure of trauma exposure: the Traumatic Life Events Questionnaire. Psychol Assess. 2000 Jun;12(2):210-24. doi: 10.1037//1040-3590.12.2.210. PMID 10887767
- [Background] Rosa AR, Sanchez-Moreno J, Martinez-Aran A, Salamero M, Torrent C, Reinares M, Comes M, Colom F, Van Riel W, Ayuso-Mateos JL, Kapczinski F, Vieta E. Validity and reliability of the Functioning Assessment Short Test (FAST) in bipolar disorder. Clin Pract Epidemiol Ment Health. 2007 Jun 7;3:5. doi: 10.1186/1745-0179-3-5. PMID 17555558
- [Background] Meyer TD, Hautzinger M. Cognitive behaviour therapy and supportive therapy for bipolar disorders: relapse rates for treatment period and 2-year follow-up. Psychol Med. 2012 Jul;42(7):1429-39. doi: 10.1017/S0033291711002522. Epub 2011 Nov 21. PMID 22099722
- [Background] Chambless DL, Hollon SD. Defining empirically supported therapies. J Consult Clin Psychol. 1998 Feb;66(1):7-18. doi: 10.1037//0022-006x.66.1.7. PMID 9489259
- [Derived] Hogg B, Valiente-Gomez A, Redolar-Ripoll D, Gardoki-Souto I, Fontana-McNally M, Lupo W, Jimenez E, Madre M, Blanco-Presas L, Reinares M, Cortizo R, Masso-Rodriguez A, Castano J, Argila I, Castro-Rodriguez JI, Comes M, Donate M, Herreria E, Macias C, Mur E, Novo P, Rosa AR, Vieta E, Radua J, Padberg F, Perez-Sola V, Moreno-Alcazar A, Amann BL. High incidence of PTSD diagnosis and trauma-related symptoms in a trauma exposed bipolar I and II sample. Front Psychiatry. 2022 Oct 20;13:931374. doi: 10.3389/fpsyt.2022.931374. eCollection 2022. PMID 36339849
- [Derived] Moreno-Alcazar A, Radua J, Landin-Romero R, Blanco L, Madre M, Reinares M, Comes M, Jimenez E, Crespo JM, Vieta E, Perez V, Novo P, Donate M, Cortizo R, Valiente-Gomez A, Lupo W, McKenna PJ, Pomarol-Clotet E, Amann BL. Eye movement desensitization and reprocessing therapy versus supportive therapy in affective relapse prevention in bipolar patients with a history of trauma: study protocol for a randomized controlled trial. Trials. 2017 Apr 4;18(1):160. doi: 10.1186/s13063-017-1910-y. PMID 28376919